CLINICAL TRIAL: NCT02120222
Title: A Phase 1 Expansion Cohort Evaluating the Selective Inhibitor of Nuclear Export (SINE) KPT-330 in Patients With Unresectable Melanoma
Brief Title: Evaluating SINE KPT-330 in Treating Patients With Melanoma That Cannot Be Removed By Surgery
Acronym: KPT-330
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kari Kendra (Other)
Collaborators: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor-Investigator, Kari Kendra, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-13124; NCI-2014-00676 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2014-04-17; First posted 2014-04-22 (Estimated); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Recurrent Melanoma
Keywords: melanoma
MeSH Terms: conditions — Melanoma | interventions — selinexor; Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (selinexor) (Experimental): Patients receive selinexor PO BIW. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity. Blood will be collected for correlative studies to perform pK (pharmacokinetics) and pDn (pharmacodynamics) analysis pretreatment on day 1 and 8 hours after treatment, on day 1 of cycles 1 and 2.
  Interventions: Drug: selinexor; Other: Correlative studies

INTERVENTIONS:
Drug: selinexor — Given PO
  Other Names: CRM1 nuclear export inhibitor KPT-330; KPT-330; selective inhibitor of nuclear export KPT-330; SINE KPT-330
Other: Correlative studies — Blood will be collected for pK and pDn analysis pretreatment on day 1 and 8 hours after treatment, on day 1 of cycles 1 and 2.
  Other Names: pharmacological studies; pharmacokinetics; pharmacodynamics

SUMMARY:
This phase I clinical trial studies the side effects of selinexor in treating patients with melanoma that cannot be removed by surgery. Drugs used in chemotherapy, such as selinexor, may stop the growth of tumor cells, by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate safety of KPT-330 (selinexor) in patients with melanoma at the maximum tolerated dose (MTD) defined by the phase 1 study.

SECONDARY OBJECTIVES:

I. To determine the clinical benefit rate (CBR) (complete response, partial response, and stable disease) of patients with unresectable melanoma.

II. To assess the efficacy at the MTD as measured by progression free survival (PFS) in patients with melanoma.

TERTIARY OBJECTIVES:

I. To validate nuclear transport inhibition resulting from treatment. II. To assess if v-raf murine sarcoma viral oncogene homolog B1 (BRAF), neuroblastoma RAS viral (v-ras) oncogene homolog (NRAS), or platelet-derived growth factor receptor, beta polypeptide (PDGFRB) mutational status impacts response.

III. To assess alteration in signaling pathways as a result of therapy with KPT-330.

IV. To assess immunologic changes resulting from treatment with KPT-330.

OUTLINE:

Patients receive selinexor orally (PO) twice weekly (BIW). Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 1 year

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent in accordance with federal, local, and institutional guidelines
* Patients with unresectable melanoma
* Patients must have received a biologic therapy (e.g. interleukin 2) and a BRAF and/or MEK inhibitor (if tumor contains the V600E or V600K mutation) for 628 metastatic disease. If patient did not receive such agents, rationale for not treating the patients with the 629 agent must be cleared with the study PI (ie no V600e/k BRAF mutation or patient with autoimmunity, thus 630 not eligible for biologic therapy).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Total white blood cell (WBC) count >= 3000/mm^3
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelet count >= 100,000/mm^3
* Bilirubin < 2 times the upper limit of normal (ULN) (except patients with Gilbert's syndrome who must have a total bilirubin of < 3 times ULN)
* Alanine aminotransferase (ALT) < 2.5 times ULN; in the case of known (radiological and/or biopsy documented) liver metastasis, ALT < 5.0 times ULN is acceptable
* Estimated creatinine clearance of >= 50 mL/min, calculated using the formula of Cockroft and Gault
* Female patients of child-bearing potential must agree to use dual methods of contraception and have a negative serum pregnancy test at screening, and male patients must use an effective barrier method of contraception if sexually active with a female of child-bearing potential; acceptable methods of contraception are condoms with contraceptive foam, oral, implantable or injectable contraceptives, contraceptive patch, intrauterine device, diaphragm with spermicidal gel, or a sexual partner who is surgically sterilized or post-menopausal; for both male and female patients, effective methods of contraception must be used throughout the study and for three months following the last dose

Exclusion Criteria:

* Patients who are pregnant or lactating
* Radiation, chemotherapy, immunotherapy or any other systemic anticancer therapy =< 2 weeks prior to initiation of therapy
* Major surgery within four weeks before initiation of therapy
* Unstable cardiovascular function:

  * Symptomatic ischemia, or
  * Uncontrolled clinically significant conduction abnormalities (e.g.: ventricular tachycardia on antiarrhythmics are excluded and 1st degree atrioventricular (AV) block or asymptomatic left anterior fascicular block [LAFB]/right bundle branch block [RBBB] will not be excluded)
  * Congestive heart failure (CHF) of New York Heart Association (NYHA) class >= 3, or
  * Myocardial infarction (MI) within 3 months of initiation of therapy
* Uncontrolled active infection within one week prior to first dose
* Known to be human immunodeficiency virus (HIV) seropositive
* Known active hepatitis A, B, or C infection; or known to be positive for hepatitis C virus (HCV) ribonucleic acid (RNA) or HBsAg (hepatitis B virus [HBV] surface antigen)
* Patients with active central nervous system (CNS) malignancy

  * Asymptomatic small lesions are not considered active
  * Treated lesions may be considered inactive if the patient is able to taper off steriods without any recurrent neurologic symptoms.
* Patients will be excluded if they have had a major resection of the bowel that could influence absorption, inflammatory bowel disease, or other gastrointestinal conditions with increased risk of perforation, history of abdominal fistula, gastrointestinal perforation within 28 days prior to beginning study treatment
* Grade >= 2 peripheral neuropathy within 14 days prior to initiation of therapy
* History of seizures, movement disorders or cerebrovascular accident within the past 5 years
* Patients with known macular degeneration or uncontrolled glaucoma
* In the opinion of the investigator, patients who are significantly below their ideal body weight
* Serious psychiatric or medical conditions that could interfere with treatment
* Participation in an investigational anti-cancer study within 3 weeks prior to initiation of therapy
* Concurrent therapy with approved or investigational anticancer therapeutic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-08-22 (Actual); Primary Completion 2018-04-08 (Actual); Study Completion 2018-04-08 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events graded using the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03 | 28 days
  Types of toxicities, incidences and severity will be summarized by descriptive statistics such as frequencies/proportions.

SECONDARY OUTCOMES:
CBR (complete response, partial response, stable disease or stable disease) using Response Evaluation Criteria in Solid Tumors | Up to 1 year
PFS | From date of registration to date of first documentation of progression or symptomatic deterioration or death due to any cause or last contact, assessed up to 1 year
  Kaplan-Meier method will be used to assess the PFS.
Change in tumor markers by immunohistochemistry | Baseline to up to 1 year
  Markers with continuous numerical data will be analyzed using linear mixed effects models (LMEMs). Binary markers (presence vs. absence) will be summarized by proportions and the confidence intervals will be calculated. Marker changes by mutation groups in plots will be presented. To correlate the marker changes with response, mainly summary statistics and plots will be used given the potentially small subgroups.

CONTACTS AND LOCATIONS:
Overall Officials: Kari Kendra, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu